CLINICAL TRIAL: NCT04882826
Title: Randomized Crossover 2 Period Single Dose Bioequivalence Study of 2 Formulations Sildenafil Tablets 100mg (Pharmtechnology LLC, Belarus) and Viagra® Tablets 100mg (Fareva Amboise, France) in Healthy Male Volunteers Under Fasting Conditions
Brief Title: Bioequivalence Study of Two Formulations of Sildenafil Tablet 100 mg in Healthy Male Volunteers Under Fasting Conditions
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Pharmtechnology LLC (Industry)
Collaborators: ClinPharmInvest, LLC (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Other
Other Study IDs: SLDF-2020-CPI-FRMT
Record Dates: First submitted 2021-05-06; First posted 2021-05-12 (Actual); Last update posted 2021-05-12 (Actual); Status verified 2021-05

CONDITIONS: Bioequivalence
Keywords: Sildenafil; Bioequivalence; Viagra

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sequence TR (Other): 22 subjects assigned to the sequence TR will receive a single 100 mg dose of the test product Sildenafil (1 x 100 mg tablet), marked as T in the sequence, in Period 1 and a single 100 mg dose of the reference product Viagra® (1 x 100 mg tablet), marked as R in the sequence, in period 2. These treatments will be administered orally with approximately 200 mL of water, in the morning, following a 10-hour overnight fast. The tablet must be swallowed whole and must not be chewed or broken.
  Interventions: Drug: Sildenafil film-coated tablet 100 mg; Drug: Viagra® film-coated tablet 100 mg
- Sequence RT (Other): 22 subjects assigned to the sequence RT will receive a single 100 mg dose of the reference product Viagra® (1 x 100 mg tablet), marked as R in the sequence, in Period 1 and a single 100 mg dose of the test product Sildenafil (1 x 100 mg tablet), marked as T in the sequence, in period 2. These treatments will be administered orally with approximately 200 mL of water, in the morning, following a 10-hour overnight fast. The tablet must be swallowed whole and must not be chewed or broken.
  Interventions: Drug: Sildenafil film-coated tablet 100 mg; Drug: Viagra® film-coated tablet 100 mg

INTERVENTIONS:
Drug: Sildenafil film-coated tablet 100 mg — Sildenafil is manufactured by Pharmtechnology LLC, Belarus. Each tablet contains 100 mg of sildenafil.
  Other Names: The test product
Drug: Viagra® film-coated tablet 100 mg — Viagra® is manufactured by Fareva Amboise, France. Each tablet contains 100 mg of sildenafil.
  Other Names: The reference product

SUMMARY:
This is an open-labeled (laboratory blinded), randomized, two period, single-center, crossover, comparative study, where each participant will be randomly assigned to the reference (Viagra®, 100 mg film-coated tablets) or the test (Sildenafil, 100 mg film-coated tablets) formulation in each period of study (sequences Test-Reference (TR) or Reference-Test (RT)), in order to evaluate if both formulations are bioequivalent

ELIGIBILITY:
Inclusion Criteria:

1. Healthy caucasian men aged between 18 to 45 years
2. The written consent of the volunteer to be included in the study
3. Verified diagnosis "healthy" according to the anamnesis data and the results of standard clinical, laboratory and instrumental examination methods, physical examination and anamnestic examination
4. Body mass index 18.5-30 kg/m² according to Quetelet's weight-height index
5. The results of an X-ray or fluorographic examination of the chest organs within the normal range (the results of an examination carried out within 12 months before the start of the study may be provided)
6. Absence of ophthalmological disease according to the data of the ophthalmological examination
7. Consent to use a double barrier method of contraception (condom + spermicide) or sexual continence, as well as consent not to take part in sperm donation from the moment of taking the drug in the first period, during the entire study and within 14 days after taking the drug in the second period research
8. Subjects are able to understand the requirements of the study, to sign a written informed consent, and also to accept all the restrictions imposed during the course of the study, and to agree to return for the required investigations

Exclusion Criteria:

1. Burdened allergic history, hypersensitivity to sildenafil or excipients that are part of any of the investigational drugs, or intolerance to these components.
2. Lactose intolerance, lactase deficiency, glucose-galactose malabsorption.
3. Anatomical deformation of penis (angulation, cavernous fibrosis, or Peyronie's disease).
4. History of priapism.
5. Hereditary retinitis pigmentosa.
6. Episodes of development of anterior non-arteritis ischemic neuropathy of the optic nerve.
7. Organic brain damage, a history of increased convulsive readiness.
8. Acute or chronic diseases of the cardiovascular, bronchopulmonary, neuroendocrine systems, and also diseases of the gastrointestinal tract, liver, kidneys and blood, eye disease.
9. Other diseases that, in the opinion of the researcher, may affect the absorption, distribution, metabolism or excretion of both drugs, or increase the risk of negative consequences for the volunteer.
10. The presence of mental disorders, including a history.
11. Surgical interventions on the gastrointestinal tract, with the exception of appendectomy.
12. Acute infectious diseases that ended less than 4 weeks before taking the drug in the first period.
13. Dehydration due to diarrhea, vomiting or other reason within the last 24 hours before taking the drug in the first period of the study, if vomiting or diarrhea wasn't a manifestation of an infectious disease.
14. Clinically significant abnormalities on the ECG, the level of systolic blood pressure (SBP) measured in the sitting position at the time of screening <100 mm Hg or ≥ 130 mm Hg and / or diastolic blood pressure (DBP) <60 mm Hg or ≥ 85 mm Hg.
15. Heart rate less than 60 beats/min or more than 90 beats/min at the time of screening, respiratory rate less than 14 or more than 18 per minute at the time of screening, body temperature below 36.0 ° C or above 37.0 °C at the time of screening.
16. Use of any prescription and OTC drugs including herbs and food additives, vitamins that can have a significant effect on the PK of sildenafil or data on the effect of which on the pharmacokinetics of sildenafil are unknown, as well as question the characterization of the volunteer as healthy, less than 14 days before taking the drug in the first period;
17. Use of well-known inhibitors or inducers of liver microsomal enzymes (barbiturates, omeprazole, cimetidine, etc.) or antiviral drugs less than 2 months before enrollment in the study.
18. The use of donors of nitric oxide, organic nitrates or nitrites in any form less than 30 days before taking of the drug in the first period.
19. Donation of plasma or blood (450 ml or more) less than 2 months (60 days) before taking the drug in the first period.
20. Consumption of caffeine and xanthine-containing drinks and products (tea, coffee, chocolate, cola, etc.), products containing poppy seeds, less than 48 hours before taking the drug in the first period.
21. Consumption of alcohol and alcohol-containing foods and beverages less than 48 hours before taking the drug in the first period.
22. Use of citrus fruits (including grapefruit and grapefruit juice) and cranberries (including juices, fruit drinks, etc.) less than 7 days before taking the drug in the first period.
23. Intake of more than 10 units alcohol per week (1 unit of alcohol is equivalent to 500 ml of beer, 200 ml of dry wine or 50 ml of spirits) or history of alcoholism, drug addiction, drug abuse.
24. Intense physical activity less than 24 hours before taking the drug in the first period.
25. Smoking more than 10 cigarettes less than 24 hours before taking the drug in the first period.
26. Participation in other clinical trials of drugs less than 3 months before taking the drug in the first period.
27. Following any low sodium diet within 2 weeks prior to study initiation, or following a special diet (vegetarian, vegan, with limited salt intake) or lifestyle (night work, extreme physical activity).
28. Test positive for syphilis, hepatitis B, hepatitis C or HIV at the time of screening.
29. Positive test for alcohol in exhaled air at screening.
30. Positive urinalysis for the content of narcotic and potent substances during screening (opiates, morphine, barbiturates, benzodiazepines, cannabinoids/marijuana).
31. The value of standard laboratory and instrumental parameters that go beyond the reference values.
32. Lack of intention of volunteers to comply with the Protocol requirements throughout the course of the study and/or lack, in the opinion of the Investigator, of the volunteers' ability to understand and evaluate the information on this study as part of the informed consent form signing process, in particular regarding the expected risks and possible discomfort.
33. Mental, physical and other reasons that do not allow the volunteer to adequately assess their behavior and correctly comply with the conditions of the research protocol.
34. Tattooing and piercing within 30 days prior to first drug administration.
35. Difficulty swallowing tablets.
36. Difficulty with taking blood (for example, difficult access to the veins).

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 44 (Estimated)
Dates: Start 2021-05-10 (Estimated); Primary Completion 2021-05-30 (Estimated); Study Completion 2021-05-30 (Estimated)

PRIMARY OUTCOMES:
Cmax of sildenafil and N-Desmethyl Sildenafil in plasma after administration of the test and the reference products. | Time points 0.00 (prior to each drug administration) and 0.17, 0.33, 0.50, 0.67, 0.83, 1.00, 1.25, 1.50, 1.75, 2.00, 2.33, 2.67, 3.00, 3.50, 4.00, 5.00, 6.00, 8.00, 10.00, 12.00, 16.00, 24.00 hours after each drug administration.
  Maximum observed concentration in plasma.
AUC0-t of sildenafil and N-Desmethyl Sildenafil in plasma after administration of the test and the reference. | Time points 0.00 (prior to each drug administration) and 0.17, 0.33, 0.50, 0.67, 0.83, 1.00, 1.25, 1.50, 1.75, 2.00, 2.33, 2.67, 3.00, 3.50, 4.00, 5.00, 6.00, 8.00, 10.00, 12.00, 16.00, 24.00 hours after each drug administration.
  Cumulative area under the concentration time curve calculated from 0 to time of last observed quantifiable concentration (TLQC) using the linear trapezoidal method

SECONDARY OUTCOMES:
Tmax of sildenafil and N-Desmethyl Sildenafil in plasma after administration of the test and the reference products. | Time points 0.00 (prior to each drug administration) and 0.17, 0.33, 0.50, 0.67, 0.83, 1.00, 1.25, 1.50, 1.75, 2.00, 2.33, 2.67, 3.00, 3.50, 4.00, 5.00, 6.00, 8.00, 10.00, 12.00, 16.00, 24.00 hours after each drug administration.
  Time of maximum observed concentration; if it occurs at more than one time point, Tmax is defined as the first time point with this value.
TLQC of sildenafil and N-Desmethyl Sildenafil in plasma after administration of the test and the reference products. | Time points 0.00 (prior to each drug administration) and 0.17, 0.33, 0.50, 0.67, 0.83, 1.00, 1.25, 1.50, 1.75, 2.00, 2.33, 2.67, 3.00, 3.50, 4.00, 5.00, 6.00, 8.00, 10.00, 12.00, 16.00, 24.00 hours after each drug administration.
  Time of last observed quantifiable concentration.
AUC0-INF of sildenafil and N-Desmethyl Sildenafil in plasma after administration of the test and the reference products. | Time points 0.00 (prior to each drug administration) and 0.17, 0.33, 0.50, 0.67, 0.83, 1.00, 1.25, 1.50, 1.75, 2.00, 2.33, 2.67, 3.00, 3.50, 4.00, 5.00, 6.00, 8.00, 10.00, 12.00, 16.00, 24.00 hours after each drug administration.
  Area under the concentration time curve extrapolated to infinity, calculated as AUC0-t + ĈLQC (the predicted concentration at time TLQC) / λZ (apparent elimination rate constant).
Residual area of sildenafil and N-Desmethyl Sildenafil in plasma after administration of the test and the reference products. | Time points 0.00 (prior to each drug administration) and 0.17, 0.33, 0.50, 0.67, 0.83, 1.00, 1.25, 1.50, 1.75, 2.00, 2.33, 2.67, 3.00, 3.50, 4.00, 5.00, 6.00, 8.00, 10.00, 12.00, 16.00, 24.00 hours after each drug administration.
  Extrapolated area (i.e. percentage of AUC0-INF due to extrapolation from TLQC to infinity).
Time point where the log-linear elimination phase begins (TLIN) of sildenafil and N-Desmethyl Sildenafil in plasma after administration of the test and the reference. products. | Time points 0.00 (prior to each drug administration) and 0.17, 0.33, 0.50, 0.67, 0.83, 1.00, 1.25, 1.50, 1.75, 2.00, 2.33, 2.67, 3.00, 3.50, 4.00, 5.00, 6.00, 8.00, 10.00, 12.00, 16.00, 24.00 hours after each drug administration.
  Time point where the log-linear elimination phase begins.
λZ of sildenafil and N-Desmethyl Sildenafil in plasma after administration of the test and the reference products. | Time points 0.00 (prior to each drug administration) and 0.17, 0.33, 0.50, 0.67, 0.83, 1.00, 1.25, 1.50, 1.75, 2.00, 2.33, 2.67, 3.00, 3.50, 4.00, 5.00, 6.00, 8.00, 10.00, 12.00, 16.00, 24.00 hours after each drug administration.
  Apparent elimination rate constant, estimated by linear regression of the terminal linear portion of the log concentration versus time curve.
Terminal elimination half-life (Thalf) of sildenafil and N-Desmethyl Sildenafil in plasma after administration of the test and the reference products. | Time points 0.00 (prior to each drug administration) and 0.17, 0.33, 0.50, 0.67, 0.83, 1.00, 1.25, 1.50, 1.75, 2.00, 2.33, 2.67, 3.00, 3.50, 4.00, 5.00, 6.00, 8.00, 10.00, 12.00, 16.00, 24.00 hours after each drug administration.
  Terminal elimination half-life, calculated as ln(2)/λZ.
Number of treatment-emergent adverse events for the test and the reference products. | Time points 0.00 (prior to each drug administration) and 0.17, 0.33, 0.50, 0.67, 0.83, 1.00, 1.25, 1.50, 1.75, 2.00, 2.33, 2.67, 3.00, 3.50, 4.00, 5.00, 6.00, 8.00, 10.00, 12.00, 16.00, 24.00 hours after each drug administration.
  The safety population will include all subjects who received at least one dose of the test or the reference product. Any significant changes will be recorded as treatment-emergent adverse events only if they are judged clinically significant by the qualified investigator or delegate.

CONTACTS AND LOCATIONS:
Overall Officials: Alexander Khokhlov, Principal Investigator — ClinPharmInvest, LLC
Locations (1):
- Private healthcare institution "Clinical Hospital "RZD-Medicine" of the city of Yaroslavl", Yaroslavl, Russia